CLINICAL TRIAL: NCT05601258
Title: Association Between Pancreatic Lipase Levels and Coronavirus Disease 2019
Brief Title: Lipase Levels and Coronavirus Disease 2019
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Cevdet Duran, Cevdet Duran, Uşak University
Other Study IDs: UsakUCevdet3
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pancreatitis; Lipase Increased
MeSH Terms: conditions — Pancreatitis | interventions — Aging; Sex; Hospitalization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with higher lipase level: patients with higher lipase levels (higher than the laboratory upper limits) in the course of SARS-CoV-2 infection
  Interventions: Other: Age, gender, hospitalization and mortality rates will be compared
- Control: patients with normal lipase levels in the course of SARS-CoV-2 infection
  Interventions: Other: Age, gender, hospitalization and mortality rates will be compared

INTERVENTIONS:
Other: Age, gender, hospitalization and mortality rates will be compared — Age, gender, hospitalization and mortality rates will be compared

SUMMARY:
Although COVID-19 disease due to Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) affects the respiratory tract, heart and coagulation system, symptoms of gastrointestinal system involvement such as abdominal pain, nausea, vomiting and diarrhea are also common.

In this study, it was aimed retrospective analysis of clinical and laboratory data of patients who developed pancreatic injury and acute pancreatitis in the course of COVID 19 disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lipase levels measured during COVID-19

Exclusion Criteria:

Patients with age <18 years Patients with pregnancy Patients whose lipase levels were not measured in the course of COVID-19 Patients with known solid organ malignacy Patients with known hematologic malignacy

Age Groups: Child, Adult, Older Adult
Study Population: Eighteen years of age or older, whose lipase level is measured in the course of COVID 19, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
The frequency of lipase enzyme elevation will be compared | From 31th March 2020 until 9th July 2021
The mortaliy rate will be compared | From 31th March 2020 until 9th July 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Cevdet Duran, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No